CLINICAL TRIAL: NCT05146609
Title: Acceptance of Hepatitis C Screening by Self-testing in High Risk and General Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Medical Doctor, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TGSS_EXCAD_AP
Record Dates: First submitted 2021-10-25; First posted 2021-12-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HR-HOSPITAL (Experimental): Patients assigned to the strategy HR-HOSPITAL, who are high risk population (HR), will receive an invitation letter for HCV screening with DBS to be performed by themselves or at the referral hospital.
  Interventions: Behavioral: Screening HCV. HR-HOSPITAL
- HR-DDP (Experimental): Patients assigned to the strategy HR-DDP, who are high risk population, will receive an invitation letter for HCV screening with DBS to be performed by themselves or at the drug dependence center (DDP) the participants used to attend.
  Interventions: Behavioral: Screening HCV. HR-DDP
- GP-HOSPITAL (Experimental): Patients assigned to the strategy GP-HOSPITAL, who are general population (GP), will receive an invitation letter for HCV screening with DBS to be performed by themselves or at the referral hospital.
  Interventions: Behavioral: Screening HCV. GP-HOSPITAL
- GP-PCC (Experimental): Patients assigned to the strategy GP-PCC, who are general population (GP), will receive an invitation letter for HCV screening with DBS to be performed by themselves or at the primary care center (PCC) to be performed by the general practitioner.
  Interventions: Behavioral: Screening HCV. GP-PCC

INTERVENTIONS:
Behavioral: Screening HCV. HR-HOSPITAL — Screening HCV in high risk population by themselves or at referral hospital.
  Arms: HR-HOSPITAL
Behavioral: Screening HCV. HR-DDP — Screening HCV in high risk population by themselves or at drug dependence center.
  Arms: HR-DDP
Behavioral: Screening HCV. GP-HOSPITAL — Screening HCV in general population by themselves or at referral hospital.
  Arms: GP-HOSPITAL
Behavioral: Screening HCV. GP-PCC — Screening HCV in general population by themselves or at primary care center.
  Arms: GP-PCC

SUMMARY:
The main purpose of the study is to evaluate the acceptance and viability of self-testing using dried blood spot (DBS) testing assisted by center of origin or referral hospital, as a strategy for screening for hepatitis C virus (HCV) in high risk population (ex-users of drug dependence centers) compared to the general population assisted by primary care centers.

DETAILED DESCRIPTION:
This is a randomized clinical trial involving patients who between 2013 and 2017 have contacted the drug dependence center and patients from general population.

After selecting those who do not meet any exclusion criteria, a letter will be sent to them inviting them to participate in this study. This letter will contain the study information sheet and informed consent, and a self-testing kit with an explanatory leaflet so that each person can carry out the test in a simple and easy way.

The main purpose of the study is to evaluate the acceptance and viability of self-testing using dried blood spot (DBS) testing, to study whether support improves participation and to identify predictors of participation.

For the present study, assuming an increase of 18% participation (from 18% to 28% offering support by the patient's referral center, and based on a previous study in our environment of self-testing in the general population), taking into account a power of 80%, alpha error of 5%, and losses of 20%, will require 346 patients per group.

ELIGIBILITY:
Inclusion criteria:

* All subjects who have contacted a drug dependence center between 2013 and 2017, as well as patients from a group of a primary care center.
* Signed informed consent.

Exclusion criteria:

* Patient's refusal to participate in the study.
* Negative HCV serology or viral load in the last year.
* Death.
* Belonging to another health area
* Not having the patient's address in the hospital's computer system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1384 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the intervention | 12 months
  Overall screening rate

SECONDARY OUTCOMES:
Viability | 12 months
  The investigators will measure and report the amount of DBS received from the participants, taking into account the group to which the participants belong.
Participation | 12 months
  Number of participants by sending their DBS and different possible factors associated to a higher rate of participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for Study of Liver. EASL Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2014 Feb;60(2):392-420. doi: 10.1016/j.jhep.2013.11.003. Epub 2013 Dec 9. No abstract available. PMID 24331294
- [Background] Baumert TF, Juhling F, Ono A, Hoshida Y. Hepatitis C-related hepatocellular carcinoma in the era of new generation antivirals. BMC Med. 2017 Mar 14;15(1):52. doi: 10.1186/s12916-017-0815-7. PMID 28288626
- [Background] Westbrook RH, Dusheiko G. Natural history of hepatitis C. J Hepatol. 2014 Nov;61(1 Suppl):S58-68. doi: 10.1016/j.jhep.2014.07.012. Epub 2014 Nov 3. PMID 25443346
- [Background] Sarin SK, Kumar M. Natural history of HCV infection. Hepatol Int. 2012 Oct;6(4):684-95. doi: 10.1007/s12072-012-9355-6. Epub 2012 Mar 9. PMID 26201520
- [Background] Buti M, Dominguez-Hernandez R, Casado MA, Sabater E, Esteban R. Healthcare value of implementing hepatitis C screening in the adult general population in Spain. PLoS One. 2018 Nov 28;13(11):e0208036. doi: 10.1371/journal.pone.0208036. eCollection 2018. PMID 30485377
- [Background] Juanbeltz R, Perez-Garcia A, Aguinaga A, Martinez-Baz I, Casado I, Burgui C, Goni-Esarte S, Reparaz J, Zozaya JM, San Miguel R, Ezpeleta C, Castilla J; EIPT-VHC Study Group. Progress in the elimination of hepatitis C virus infection: A population-based cohort study in Spain. PLoS One. 2018 Dec 4;13(12):e0208554. doi: 10.1371/journal.pone.0208554. eCollection 2018. PMID 30513107
- [Background] Morales-Arraez D, Hernandez-Guerra M. Electronic Alerts as a Simple Method for Amplifying the Yield of Hepatitis C Virus Infection Screening and Diagnosis. Am J Gastroenterol. 2020 Jan;115(1):9-12. doi: 10.14309/ajg.0000000000000487. No abstract available. PMID 31833860
- [Background] Fitz JG. Hepatology after Hepatitis C. Dig Dis. 2016;34(5):603-6. doi: 10.1159/000445276. Epub 2016 Jun 22. PMID 27332966
- [Background] Crespo J, Albillos A, Buti M, Calleja JL, Garcia-Samaniego J, Hernandez-Guerra M, Serrano T, Turnes J, Acin E, Berenguer J, Berenguer M, Colom J, Fernandez I, Fernandez Rodriguez C, Forns X, Garcia F, Rafael Granados, Lazarus JV, Molero JM, Molina E, Perez Escanilla F, Pineda JA, Rodriguez M, Romero M, Roncero C, Saiz de la Hoya P, Sanchez Antolin G. Elimination of hepatitis C. Positioning document of the Spanish Association for the Study of the Liver (AEEH). Gastroenterol Hepatol. 2019 Nov;42(9):579-592. doi: 10.1016/j.gastrohep.2019.09.002. Epub 2019 Oct 5. English, Spanish. PMID 31594683
- [Background] Morales-Arraez D, Hernandez-Bustabad A, Medina-Alonso MJ, Santiago-Gutierrez LG, Garcia-Gil S, Diaz-Flores F, Perez-Perez V, Nazco J, Fernandez de Rota Martin P, Gutierrez F, Hernandez-Guerra M. Telemedicine and decentralized hepatitis C treatment as a strategy to enhance retention in care among people attending drug treatment centres. Int J Drug Policy. 2021 Aug;94:103235. doi: 10.1016/j.drugpo.2021.103235. Epub 2021 Apr 7. PMID 33838399
- [Background] Bedford J, Enria D, Giesecke J, Heymann DL, Ihekweazu C, Kobinger G, Lane HC, Memish Z, Oh MD, Sall AA, Schuchat A, Ungchusak K, Wieler LH; WHO Strategic and Technical Advisory Group for Infectious Hazards. COVID-19: towards controlling of a pandemic. Lancet. 2020 Mar 28;395(10229):1015-1018. doi: 10.1016/S0140-6736(20)30673-5. Epub 2020 Mar 17. No abstract available. PMID 32197103
- [Background] Blach S, Kondili LA, Aghemo A, Cai Z, Dugan E, Estes C, Gamkrelidze I, Ma S, Pawlotsky JM, Razavi-Shearer D, Razavi H, Waked I, Zeuzem S, Craxi A. Impact of COVID-19 on global HCV elimination efforts. J Hepatol. 2021 Jan;74(1):31-36. doi: 10.1016/j.jhep.2020.07.042. Epub 2020 Aug 7. PMID 32777322